CLINICAL TRIAL: NCT04459559
Title: Usability Study of a Novel Tactile Cueing Device for Patients With Parkinson's Disease: A Monocentric Interventional Study
Brief Title: Usability of a Novel Cueing Device for Patients With Parkinson's Disease
Acronym: TCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Rehaklinik Zihlschlacht AG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZS_01_2020
Record Dates: First submitted 2020-06-11; First posted 2020-07-07 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Freezing of Gait; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The proposed trial is designed as an explorative, open label, non-randomised, uncontrolled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Using the Tactile Cueing Device
  Interventions: Device: Tactile Cueing Device

INTERVENTIONS:
Device: Tactile Cueing Device — Each participant receives an individual training on how to use the Tactile Cueing Device and the set-up of the TCD will be done according to the results of a 10MWT and the participant's preferences. Gait assessments with an activated or deactivated TCD are executed using the Timed Up and Go test, the 2-Minute Waling test and a treadmill (C-Mill). Also a long-term test run of the TCD during one day is planned.

SUMMARY:
Hypokinetic gait disorder and Freezing of Gait (FOG) are frequent symptoms in the advanced stage of Parkinson's disease (PD). These impair quality of life and significantly increase the risk of falls. External movement pacemakers have been developed to improve gait and avert FOG by cueing strategies. The investigators developed a smart, small and lightweight, easy-to-handle wearable tactile cueing device (TCD), consisting of a control unit, two pulse generators and a battery-driven power supply. The device is programmed via a Graphical User Interface (GUI).

ELIGIBILITY:
Inclusion Criteria:

* Include patients who suffer from advanced PD. Characteristic symptoms of parkinsonian gait like hypokinetic movements and/or FOG have to be present.
* Parkinsonian gait is measured by the following items of the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS): item 2.12, item 2.13, item 3.10 and item 3.11. The Hoehn and Yahr (HY) stage during ON is 1-4/5.
* MoCA ≥ 22/30.
* Participant has signed the informed consent.

Exclusion Criteria:

* Inability of the participant to understand the IC or to follow the procedures of the study (as judged by the Qualified Physician).
* Significantly, impaired cognitive skills render the participant unable to use the TCD.
* Presence of severe motor fluctuations and severely impaired walking ability as defined by HY stage V during ON.
* Clinically relevant skin lesions on the wrist or fixation points (usually the thighs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Setup cueing device | 2 weeks
  Time needed for the setup [in seconds] and the variations of the different setup parameters (cueing length [seconds], cueing strength [% of maximum], cueing cadence [count/minutes]) between the days of usage. Overall descriptive summary of the variation between the different setup parameters during the days of usage.
System Usability Scale | 2 weeks
  Items defined by the System Usability Scale: 5-point Likert scale ('strongly disagree' to 'strongly agree').
Usability | 2 weeks
  Usability of the cueing device is measured by a self-developed questionnaire.
Acceptance | 2 weeks
  Acceptance is measured by a self-developed questionnaire.
Frequency using the device | 2 weeks
  How often the device is used (counts logging protocol).

SECONDARY OUTCOMES:
Walking speed [meters/second] | 1 week
  Calculated by the assessments 10 meter walk test and 2-minute walk test.
Cadence [steps/minute] | 1 week
  Number during 10 meter walk test. Also measured by a system of movement analysis (C-Mill MOTEK).
Walking distance [in meters] | 1 week
  Measured by a digital measuring wheel during 2-minute walk test. Also measured by a system of movement analysis (C-Mill MOTEK).
Step length right/left [in meters] | 1 week
  Measured by a system of movement analysis (C-Mill MOTEK).
Initial step latency [in seconds] | 1 week
  Extracted from video documentation by a blinded rater.
Number of FOG | 1 week
  Extracted from video documentation by a blinded rater.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Schweinfurther, M.A., Principal Investigator — Rehaklinik Zihlschlacht AG
Locations (1):
- Rehaklinik Zihlschlacht AG, Zihlschlacht, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachlin M, Plotnik M, Roggen D, Maidan I, Hausdorff JM, Giladi N, Troster G. Wearable assistant for Parkinson's disease patients with the freezing of gait symptom. IEEE Trans Inf Technol Biomed. 2010 Mar;14(2):436-46. doi: 10.1109/TITB.2009.2036165. Epub 2009 Nov 10. PMID 19906597
- [Background] Baker K, Rochester L, Nieuwboer A. The effect of cues on gait variability--reducing the attentional cost of walking in people with Parkinson's disease. Parkinsonism Relat Disord. 2008;14(4):314-20. doi: 10.1016/j.parkreldis.2007.09.008. Epub 2007 Nov 7. PMID 17988925
- [Background] Giladi N, Nieuwboer A. Understanding and treating freezing of gait in parkinsonism, proposed working definition, and setting the stage. Mov Disord. 2008;23 Suppl 2:S423-5. doi: 10.1002/mds.21927. No abstract available. PMID 18668629